CLINICAL TRIAL: NCT06264024
Title: Simultaneous pHototherapeutic Keratectomy and corneAl Collagen cRosslinking in Eyes With Keratoconus: a Randomized Trial (SHARK)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Olav Kristianslund, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 519516
Record Dates: First submitted 2024-01-29; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Keratoconus
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CXL (Active Comparator): Treatment with CXL alone
  Interventions: Procedure: Corneal collagen cross linking (CXL)
- CXL and t-PTK (Experimental): Treatment with t-PTK combined with CXL
  Interventions: Procedure: Corneal collagen cross linking (CXL); Procedure: Transepithelial phototherapeutic keratectomy (t-PTK)

INTERVENTIONS:
Procedure: Corneal collagen cross linking (CXL) — Use of Avedro Inc. KXL 1 system to stop progression of keratoconus
Procedure: Transepithelial phototherapeutic keratectomy (t-PTK) — Use Alcon Wavelight 500, excimer laser to remove the epithelium and some of the stroma over apex
  Arms: CXL and t-PTK

SUMMARY:
The goal of this clinical trial is to compare CXL with combined treatment with CXL and t-PTK.

The main questions it aims to answer are whether combined treatment can give better visual acuity and if the treatments are equally safe.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years or older at the time of signing the informed consent form. There is no upper age limit.
* Progressive keratoconus with indication for CXL
* Corneal thickness ≥ 420 μm

Exclusion Criteria:

* Other eye disease causing visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2034-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 month after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Risk of progression | 1 year after surgery
  Change in keratometric values

SECONDARY OUTCOMES:
Visual acuity | 3 month after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Visual acuity | 6 month after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Visual acuity | 1 year after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Visual acuity | 2 years after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Visual acuity | 5 years after surgery
  Uncorrected and corrected distance visual acuity in logMAR
Risk of progression | 1 month after surgery
  Change in keratometric values
Risk of progression | 3 months after surgery
  Change in keratometric values
Risk of progression | 6 months after surgery
  Change in keratometric values
Risk of progression | 2 years after surgery
  Change in keratometric values
Risk of progression | 5 years after surgery
  Change in keratometric values
Depth of demarcation line (OCT) | 1 month after surgery
  Measured with corneal optical coherence tomography (OCT)
Depth of demarcation line (confocal microscopy) | 1 month after surgery
  Measured with confocal microscopy
Patient reported outcome measure (PROMs) | 1 month after surgery
  National eye institute Visual Function Questionnaire 25
Patient reported outcome measure (PROMs) | 6 months after surgery
  National eye institute Visual Function Questionnaire 25
Patient reported outcome measure (PROMs) | 2 years after surgery
  National eye institute Visual Function Questionnaire 25
Patient reported pain after surgery | 48 hours after surgery
  Pain the first 48 hours after the surgery graded on visual analogue scale (VAS); 0 to 10 cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophhtalmology, University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided